CLINICAL TRIAL: NCT05473546
Title: Gastrointestinal Complications of Artificial Nutrition in ICU: a Prospective Observational Study (NUTRITI)
Brief Title: Diarrhea and Stipsis in Critically Ill Patients (NUTRITI)
Acronym: NUTRITI
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Cristian Deana, Principal Investigator, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: NUTRITI
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Critical Illness; Nutritional and Metabolic Disease; Nutritional Deficiency; ICU Acquired Weakness; Enteral Feeding Intolerance; Diarrhea; Constipation
MeSH Terms: conditions — Critical Illness; Metabolic Diseases; Malnutrition; Diarrhea; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRITICALLY ILL PATIENTS: ADULTS PATIENTS ADMITTED TO ICU DUE TO ACUTE ILLNESS THAT REQUIRE AT LEAST 72H OF STAY.
  FOR THE FIRST 7 DAYS OF STAY IN ICU, DATA ABOUT NUTRITIONAL INTERVENTION WILL BE RECORDED SUCH AS: ROUTE OF NUTRITION ADMINISTRATION, AMOUNT OF NUTRITION DELIVERED PER DAY, CALORIC TARGETS, PROTEIN REQUIREMENTS, diarrhea, CONSTIPATION, BIA ANALYSIS.
  Interventions: Other: ARTIFICIAL NUTRITION

INTERVENTIONS:
Other: ARTIFICIAL NUTRITION — ARTIFICIAL NUTRITION

SUMMARY:
This study prospectively observed the complications intended as diarrhea or sti-sis that critically ill patients developed within 7 days after ICU admission.

In addition, secondary aims investigated through bioimpedenziometry the loss of lean body mass and changes in phase angle during the same period of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* ICU ANTICIPATED LENGTH OF STAY > 72 HOURS
* AGE > 18 YEARS
* NEED FOR ARTIFICIAL NUTRITION

Exclusion Criteria:

* AGE < 18 YEARS
* ICU ANTICIPATED LENGTH OF STAY < 72 HOURS
* NO NEED FOR ARTIFICIAL NUTRITION
* BMI<16 KG/M2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ADULTS ICU CRITICALLY ILL PATIENTS REQUIRING ICU ADMISSION DUE TO ACUTE ILLNESS WITH ANTICIPATED ICU STAY > 72 HOURS AND NEEDING ARTIFICIAL NUTRITION
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
FREQUENCY OF diarrhea WITHIN 72 HOURS AFTER ICU ADMISSION | 7 DAYS
  REGISTER DIARROHEA (EMISSION OF FAECES> 200 ML IN 24 HOURS) EPISODES

SECONDARY OUTCOMES:
FREQUENCY OF CONSTIPATION WITHIN 7 DAYS AFTER ICU ADMISSION | 7 DAYS
  REGISTER CONSTIPATION EPISODES WITHIN 7 DAYS AFTER ADMISSION IN ICU
LOSS OF LEAN BODY MASS AFTER 7 DAYS IN ICU | 7 DAYS
  Loss of at least 7% of lean body mass
CHANGES IN PHASE ANGLE AFTER 7 DAYS IN ICU | 7 DAYS
  Measure of phase angle

CONTACTS AND LOCATIONS:
Overall Officials: CRISTIAN DEANA, MD, Principal Investigator — Health Integrated Agency of Friuli Centrale, via Pozzuolo 330, 33100 Udine, Italy
Locations (1):
- Cristian Deana, Udine, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Danielis M, Mattiussi E, Piani T, Iacobucci A, Tullio A, Molfino A, Vetrugno L, Deana C; Nutriti Study Group. Diarrhoea and constipation during artificial nutrition in intensive care unit: A prospective observational study. Clin Nutr ESPEN. 2023 Oct;57:375-380. doi: 10.1016/j.clnesp.2023.07.007. Epub 2023 Jul 20. PMID 37739681